CLINICAL TRIAL: NCT07031063
Title: Safety, Tolerability and Effectiveness of DOlutegravir/Lamivudine Compared With Bictegravir/Tenofovir Alafenamide/Emtricitabine in People Living With HIV Without Antiretroviral Experience (TEOTL)
Brief Title: Safety, Tolerability and Effectiveness of DTG/3TC vs BIC/TAF/FTC in PWH Without Antiretroviral Experience
Acronym: TEOTL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, José Antonio Mata Marín, Dr. José Antonio Mata Marín, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2025-3502-071
Record Dates: First submitted 2025-05-25; First posted 2025-06-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: HIV Infection; Metabolic Syndrome; Antiretroviral Treatment
Keywords: HIV; dual-therapy; BIC/TAF/FTC; DTG/3TC; metabolic syndrome
MeSH Terms: conditions — HIV Infections; Metabolic Syndrome | interventions — Dual Anti-Platelet Therapy; bictegravir; imidazole mustard; Racivir

STUDY DESIGN:
Intervention Model Description: Study design: Experimental, longitudinal, prospective, randomized 1:1, open-label.
  Study type: Open-label, randomized clinical trial. Study location: Infectious Diseases Hospital. Study duration: 144 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIC/TAF/FTC (Active Comparator): Bictegravir/ tenofovir alafenamide/ emtricitabine 50/ 25/ 200 mg. It is the usual therapy, consisting of 3 drugs in a single tablet, based on an integrase inhibitor, and 2 nucleoside analogues.
  Interventions: Drug: Bictegravir (BIC) plus Emtricitabine (FTC) plus Tenofovir Alafenamide (TAF)
- DTG/3TC (Experimental): Dolutegravir/lamivudine 50/300 mg. 2-drug therapy in 1 tablet, co-formulated with 1 integrase inhibitor and 1 nucleoside analogue
  Interventions: Drug: DTG/3TC

INTERVENTIONS:
Drug: DTG/3TC — Dual therapy of 2 drugs co-formulated in 1 tablet: Dolutegravir 50 mg/ lamivudine 300 mg, it is the experimental group
  Other Names: Dual therapy
  Arms: DTG/3TC
Drug: Bictegravir (BIC) plus Emtricitabine (FTC) plus Tenofovir Alafenamide (TAF) — It is a triple-drug antiretroviral drug co-formulated in a single tablet. It contains bictegravir 50 mg, tenofovir alafenamide 25 mg, and emtricitabine 200 mg. It is the standard therapy.
  Arms: BIC/TAF/FTC

SUMMARY:
Background: The primary goal of antiretroviral therapy is to prevent HIV-associated morbidity and mortality. The effectiveness of first-line regimens is supported by a large number of clinical trials; current concerns focus on the long-term adverse effects of antiretrovirals, especially integrase strand transfer inhibitors, as they have been associated with significant weight gain, which may be associated with increased cardiovascular risk.

Objective: To determine the effectiveness, safety, and tolerability of Dolutegravir/Lamivudine (DTG/3TC) compared with Bictegravir/Tenofovir Alafenamide/Emtricitabine (BIC/TAF/FTC) in treatment-naive people living with HIV (PWH). Materials and methods: With prior approval from the Ethics and Scientific Research Committee 3502, an open-label, randomized clinical trial will be conducted at the Infectious Diseases Hospital of the National Medical Center "La Raza" from November 2024 to May 2026. Recently diagnosed PWH with no history of PrEP and/or PeP use, without hospitalization criteria, and without a diagnosis of metabolic syndrome based on ATP-III criteria will be identified. They will be invited to participate in the study and, if they accept, they will sign an informed consent form. They will be randomized to start a BIC/TAF/FTC or DTG/3TC 1:1 regimen. Laboratory studies, vital signs, and somatometry including bioimpedance will be performed at 4, 12, 24, 36, 48, 72, 96, 120, 144 weeks of follow-up; viral load and CD4+ count will be measured at weeks 12, 24, 48, 72, 96, 120, 144 weeks after the start of treatment. Sampling will be non-probabilistic; the distribution will be identified using the Kolmogorov-Smirnoff test, and measures of central tendency and percentages will be expressed. Comparisons will be made using the Mann-Whitney U test. Qualitative data will be analyzed using the x2 or Fisher's exact test. Group analysis will be performed at 12, 24, 48, 96 and 144 weeks using the Wilcoxon test. A P value ≤0.05 with a 95% confidence interval will be considered statistically significant.

DETAILED DESCRIPTION:
With prior approval of the protocol by the Local Ethics and Scientific Research Committee 3502, PWH attending the HIV clinic at the Infectious Diseases Hospital who are ART (antiretroviral therapy) naive and meet all the protocol inclusion criteria will be identified. They will be invited to participate in the study protocol, and will sign informed consent during the medical visit. If they accept, they will be explained that they can withdraw from the study whenever they wish. The initial medical interview will then be conducted to assess the sociodemographic, clinical, and comorbid characteristics of the PWH, eating habits, exercise, alcoholism and smoking; in addition, anthropometric measurements will be taken with the 4-point bioimpedance equipment (FitScan segmental body composition monitor C-545F), which expresses weight in kilograms, water in %, muscle in kg, bone in kg, fat in %; waist and hip will be recorded on the data collection sheet. The principal or associate investigator will take measurements in centimeters, in addition to vital signs such as blood pressure, heart rate, respiratory rate, oxygen saturation, prior to entering the study. In addition, in that first consultation, the following will be assessed: Glucose, creatinine, lipid profile, liver function test, complete blood count, viral load, CD4+, hepatitis B virus serology, hepatitis C virus serology, and VDRL. Randomization will be performed using the MEDSHARING digital system for each of the two arms, consisting of DTG/3TC or BIC/FTC/TAF. Follow-up appointments will be held at 4, 12, 24, 36, 48, 72, 96, 120, 144 weeks after randomization with further laboratory studies at baseline and at 4, 12, 24, 36, 48, 72, 96, 120, 144 week. Glucose, creatinine, lipid profile, liver profile, complete blood count, adverse events by organ and system, and DAIDS scale will be assessed at 4, 12, 24, 48, 72, 96, 120, 144 weeks after randomization; HIV-1 viral load and CD4+ count will be assessed at 12, 24, 48, 72, 96, 120 and 144 weeks after study entry.Also, Neuropsychiatric disorders will be assessed with scales for depression, anxiety and insomnia: Hospital Anxiety and Depression Scale (HADS-D, HADS-A), Insomnia Severity Index (ISI), Patient Health Questionnaire (PHQ-9) prior to entering the protocol, at 4, 12, 24, 48 72, 96, 120 and 144 weeks after randomization; satisfaction with the treatment and distress associated with it will be assessed using the HIVTSQ and HIVSDM scales will be measured after 4, 12, 24, 48, 72, 96, 129, 144 weeks after randomization.

Sampling and Sample Calculation Sampling will be simple random sampling (1:1), with participation in the study offered to all ART-naive PWH who meet the selection criteria and sign the informed consent form. For this study, the target sample size was 103 participants per treatment group, based on 80% power, an α level of 2.5%, a non-inferiority margin of -10% for virologic efficacy (non-inferiority is established if the lower bound of the 2-sided 95% CI for the difference in response is greater than -10% between the two groups), and an assumed true response of 93% at week 48 for both treatment groups. Considering a 20% attrition rate, a total of 124 patients (62 PWH in each arm) are planned for enrollment.

Statistical Analysis Data will be described using proportions, frequencies, or percentages for categorical variables and using mean and standard deviation or median and percentile, according to their Kolmogorov-Smirnov distribution, for quantitative variables.

The incidence rate of metabolic syndrome, significant weight gain, dyslipidemia, overweight/obesity, and dyslipidemia will be calculated.

The Chi-square test or Fisher's exact test will be used to determine the relative risk of developing metabolic changes with the factors analyzed.

In the bivariate analysis, the paired T test or Wilcoxon paired rank sum test will be used to assess statistical significance at baseline at 48 weeks of follow-up. Statistical significance will be considered as a p value ≤0.05 with a 95% CI. For measurements at baseline, 24, and 48 weeks, the Friedman test or ANOVA will be used, depending on the type of variable.

The differences between the two groups with respect to metabolic changes and the variables studied will be determined using the Student t test or the Mann-Whitney U test, as appropriate.

In the multivariate analysis, binary logistic regression will be performed on all variables that were statistically significant in the bivariate analysis to determine the independence of the variables. Statistical analysis will be performed using SPSS (IBM) version 29.0.2 for the Mac OS Ventura operating system.

This protocol will be submitted to the institution's Ethics and Scientific Research Committee for authorization in accordance with international guidelines, including the Declaration of Helsinki, the international guidelines for biomedical ETHICS This protocol will be submitted to the institution's Ethics and Scientific Research Committee for authorization in accordance with international guidelines, including the Declaration of Helsinki, the international guidelines for biomedical research involving human subjects, from the Council for International Organizations of Medical Sciences (CIOMS) and the World Health Organization (WHO), as well as the Guidelines for Good Clinical Practice of the International Conference on Harmonization of Technical Requirements for the Registration of Pharmaceuticals for Human Use (ICH).

Confidentiality of results: This protocol will be conducted in accordance with the guidelines of local hospital authorities and based on legal structures that do not overrule the Mexican Social Security Institute. All procedures will be in accordance with the provisions of the Regulations of the General Health Law on Clinical Research. Likewise, this study will comply with the Organic Law based on public statistics, which guarantees that those providing information will be included, with the exception of identifying individuals. A unique folio number will be established on the data collection sheet, where the study will be entered, and all personal data of participants will be removed.

In the Regulations of the General Health Law on Health Research, Article 17, the randomization process considers a risk greater than minimal.

The regimens that will be used in the treatment of ART-naive PWH are recommended by national and international guidelines, so candidate PWH will receive the best treatment option in Mexico.

The probability of complications corresponding to the adverse events inherent to each treatment regimen corresponds to the adverse events inherent to each treatment regimen. Furthermore, laboratory tests are usually requested for monitoring PWH who begin ART in IMSS units. Obtaining laboratory studies may be associated with adverse events related to venipuncture and the use of sterile materials, such as pain, bruising, vascular injuries, nerve injuries, or infections. If any of these occur, participants will be instructed to seek evaluation and will receive medical treatment if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 years of age , diagnosed with HIV, and naive to antiretroviral treatment.
2. HIV-1 RNA quantified by RT-PCR ≥500 and less than 500,000 copies/mL.
3. No history of PrEP or PEP use.
4. Estimated glomerular filtration rate ≥30 mL/min/1.73 m2 SC.
5. No current or planned use of medications associated with significant weight changes during the study period.
6. Be a beneficiary of the Mexican Social Security Institute treated at the Infectious Diseases Hospital, La Raza National Medical Center.
7. Willingness of the participant to give consent.

Exclusion Criteria:

1. Diagnosis of metabolic syndrome.
2. uncontrolled diabetes
3. Contraindication to the use of INSTIs.
4. Known mutations in any of the components of either regimen (second-generation INSTIs, 3TC/FTC, or TAF).
5. Co-medications that have potential interactions with any of the components of the antiretroviral regimens.
6. Coinfection with hepatitis B or hepatitis C virus.
7. High cardiovascular risk (Framinham >20% or AHA/ACC >7.5%).
8. Use of recreational drugs with anorexigenic potential (crystal, methamphetamines, cocaine) 60 days prior to randomization.
9. Hospitalization for acute or severe illness 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine the effectiveness of Dolutegravir/Lamivudine compared with Bictegravir/Tenofovir Alafenamide/Emtricitabine in ART-naive people with HIV at 144 weeks of treatment. | 144 weeks of follow-up with interim analysis at 48 and 96 weeks
  -Effectiveness: Number of participants with viral load measurement (HIV-1 RNA) <50 copies/mL at 144 weeks of follow-up for PWH treated with DTG/3TC or BIC/FTC/TAF, expressed in proportions.
To determine the safety of Dolutegravir/Lamivudine compared with Bictegravir/Tenofovir Alafenamide/Emtricitabine in ART-naive people living with HIV at 144 weeks of treatment. | 144 weeks, with intermediate measurements at 48 and 96 weeks
  Number of participants with treatment-related adverse events as assessed of serious adverse events (WHO grade 3 or 4) for PWH treated with DTG/3TC or BIC/FTC/TAF at 144 weeks, expressed in proportions of new cases.
To determine the tolerability of Dolutegravir/Lamivudine compared with Bictegravir/Tenofovir Alafenamide/Emtricitabine in ART-naive people living with HIV at 144 weeks of treatment. | 144 weeks, intermediate measurements at 48 and 96 weeks
  Number of participants with secondary events associated with ART for PWH treated with DTG/3TC or BIC/FTC/TAF at 144 weeks expressed in proportions and percentages, graded from 1 to 4 according to DAIDS: Grade I: mild Grade II: moderate Grade III: severe Grade IV: life-threatening

SECONDARY OUTCOMES:
Metabolic syndrome incidence in DTG/3TC vs BIC/TAF/FTC at 144 weeks | 144 weeks, interim analyses at 48 and 96 weeks
  To determine the incidence of metabolic syndrome in ART-naive PWH initiating a regimen containing DTG/3TC compared with BIC/FTC/TAF after 48 weeks of follow-up, determined by the ATPIII criteria.
To evaluate changes in cardiovascular risk based on AHA/ACC score in ART-naive PWH starting a regimen with DTG/3TC compared with BIC/FTC/TAF after 144 weeks of follow-up. | 144 weeks, with interim analyses at 48 and 96 weeks
  To evaluate and compare changes in cardiovascular risk based on the ASCVD (Atherosclerotic Cardiovascular Disease) 2013 Risk Calculator from American College of Cardiology (ACC) and American Heart Association in ART-naive PWH initiating DTG/3TC regimen compared with BIC/FTC/TAF after 144 weeks of follow-up. This is classified in percentage as follows:
  High cardiovascular risk: ≥20% Borderline cardiovascular risk: ≥5%-<7.5% Low cardiovascular risk: <5% The score is directly proportional to the risk, and determines the 10-year risk of ASCVD, for example: myocardial infarction, stroke, or death due to coronary heart disease or stroke
To determine the incidence of overweight/obesity in ART-naive PWH initiating a DTG/3TC regimen compared with BIC/FTC/TAF after 144 weeks of follow-up. | 144 weeks, with interim analyses at 48 and 96 weeks
  To determine incidence of overweight/obesity by body mass index (BMI) ART-naive PWH initiating a DTG/3TC regimen compared with BIC/FTC/TAF after 144 weeks of follow-up.
To determine significant weight changes in ART-naive PWH initiating a DTG/3TC regimen compared with BIC/FTC/TAF after 144 weeks of follow-up. | 144 weeks, with interim analyses at 48 and 96 weeks
  To determine significant weight changes (>10% body weight gain) in proportions and percentages in ART-naive PWH initiating a DTG/3TC regimen compared with BIC/FTC/TAF after 144 weeks of follow-up.
To determine the incidence of virologic failure in ART-naive in PWH treated with DTG/3TC compared with BIC/TAF/FTC at 144 weeks of follow-up | 144 weeks, with intermediate measurements at 48 and 96 weeks
  The incidence of virological failure is those new cases of virological failure, defined in Mexico as 2 consecutive determinations in a period of 6 months with HIV-1 viral load >200 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: José A Mata, Master degree, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital de infectología, Centro Médico Nacional La Raza, Mexico City, Azcapotzalco, Mexico

IPD SHARING:
Plan to Share IPD: No
Participant data are confidential and may be requested from the principal investigator.

REFERENCES:
- [Background] Gallant J, Lazzarin A, Mills A, Orkin C, Podzamczer D, Tebas P, Girard PM, Brar I, Daar ES, Wohl D, Rockstroh J, Wei X, Custodio J, White K, Martin H, Cheng A, Quirk E. Bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir, abacavir, and lamivudine for initial treatment of HIV-1 infection (GS-US-380-1489): a double-blind, multicentre, phase 3, randomised controlled non-inferiority trial. Lancet. 2017 Nov 4;390(10107):2063-2072. doi: 10.1016/S0140-6736(17)32299-7. Epub 2017 Aug 31. PMID 28867497
- [Background] Durable Efficacy of Dolutegravir Plus Lamivudine in Antiretroviral Treatment-Naive Adults With HIV-1 Infection: 96-Week Results From the GEMINI-1 and GEMINI-2 Randomized Clinical Trials: Erratum. J Acquir Immune Defic Syndr. 2020 Jul 1;84(3):e21. doi: 10.1097/QAI.0000000000002394. PMID 32530908
- [Background] Cahn P, Madero JS, Arribas JR, Antinori A, Ortiz R, Clarke AE, Hung CC, Rockstroh JK, Girard PM, Sievers J, Man C, Currie A, Underwood M, Tenorio AR, Pappa K, Wynne B, Fettiplace A, Gartland M, Aboud M, Smith K; GEMINI Study Team. Dolutegravir plus lamivudine versus dolutegravir plus tenofovir disoproxil fumarate and emtricitabine in antiretroviral-naive adults with HIV-1 infection (GEMINI-1 and GEMINI-2): week 48 results from two multicentre, double-blind, randomised, non-inferiority, phase 3 trials. Lancet. 2019 Jan 12;393(10167):143-155. doi: 10.1016/S0140-6736(18)32462-0. Epub 2018 Nov 9. PMID 30420123
- [Background] Kelly SG, Nyaku AN, Taiwo BO. Two-Drug Treatment Approaches in HIV: Finally Getting Somewhere? Drugs. 2016 Apr;76(5):523-31. doi: 10.1007/s40265-016-0553-8. PMID 26886135